CLINICAL TRIAL: NCT02194153
Title: Surveillance of Patients With Suspected Acute Myocardial Infarction That Receive Prehospital or Early Inhospital (Emergency Department) Thrombolysis With Metalyse ®
Brief Title: Surveillance of Patients With Suspected Acute Myocardial Infarction That Receive Early Inhospital Thrombolysis With Metalyse
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1123.16
Record Dates: First submitted 2014-07-17; First posted 2014-07-18 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Metalyse: Metalyse weight-adjusted
  Interventions: Drug: Metalyse weight-adjusted

INTERVENTIONS:
Drug: Metalyse weight-adjusted

SUMMARY:
Obtaining data on efficacy (e.g. complete ST-segment resolution) depending on the time of treatment initiation and safety of prehospital and early hospital thrombolysis with Metalyse® in a real life setting outside clinical trials.

ELIGIBILITY:
Inclusion criteria:

* Male and female patient with suspected myocardial infarction, e.g. during transportation to the hospital by ambulance. No patient younger than 18 years.
* Possibility of obtaining relevant information concerning indication or contraindication of thrombolysis in each patient
* Typical chest pain with a duration of more than 30 minutes
* Definite infarction signs in a 12-lead-ECG with ST-elevation > 0.1 millivolt (mV) in > 2 leads or recent left bundle branch block with typical clinical signs
* Symptom onset <= 6 hours

Exclusion criteria:

* Patients older than 75 years (exception: patients appear much younger)
* Low body weight
* No persons under 18
* contraindications according to summary of product characteristics (SPC) for Metalyse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: prehospital or emergency room patients
Sampling Method: Non-Probability Sample
Enrollment: 351 (Actual)
Dates: Start 2001-05; Primary Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
Complete ST-segment resolution | up to 30 days
Pain relief | 90 min, 120 min, up to 30 days after treatment initiation
  yes/no question
Change in creatine kinase (CK) | up to 24 hours
Change in creatine kinase-MB (CK-MB) | up to 24 hours
Change in troponin | up to 24 hours